CLINICAL TRIAL: NCT06538779
Title: Sonographic Examination of Median Nerve Variations and Characteristics Observed in Healthy and Carpal Tunnel Syndrome Patients
Brief Title: Sonographic Examination of Median Nerve Variations
Status: Recruiting | Type: Observational
Sponsor: Yunus Burak Bayır (Other Government)
Responsible Party: Sponsor-Investigator, Yunus Burak Bayır, Yunus Burak Bayır, Principal İnvestigator, Ankara Etlik City Hospital
Organization: Ankara Etlik City Hospital (Other Government)
Other Study IDs: Median nerve variations
Record Dates: First submitted 2024-08-01; First posted 2024-08-06 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Carpal Tunnel Syndrome
Keywords: bifid median nerve; carpal tunnel syndrome; variations of median nerve; sonography
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- normal median nerve in carpal tunnel syndrome: Patients' general pain will be assessed with Visual Analog Scale (Global Pain), symptom severity and functional status will be assessed with Boston Carpal Tunnel Questionnaire, hand grip strength will be measured with dynamometer. Patient hand diagram will be marked according to patient's sensory symptoms. Median nerve cross-sectional area measurement at pisiform level with ultrasound, distal motor latency and sensory nerve conduction velocity with emg will be performed and recorded. Median nerve stiffness will be assessed with real-time elastography.
  Interventions: Diagnostic Test: elastography,usg
- median nerve variation in carpal tunnel syndrome: Patients' general pain will be assessed with Visual Analog Scale (Global Pain), symptom severity and functional status will be assessed with Boston Carpal Tunnel Questionnaire, hand grip strength will be measured with dynamometer. Patient hand diagram will be marked according to patient's sensory symptoms. Median nerve cross-sectional area measurement at pisiform level with ultrasound, distal motor latency and sensory nerve conduction velocity with emg will be performed and recorded. Median nerve stiffness will be assessed with real-time elastography.
  Interventions: Diagnostic Test: elastography,usg

INTERVENTIONS:
Diagnostic Test: elastography,usg — Patients' general pain will be assessed with Visual Analog Scale (Global Pain), symptom severity and functional status will be assessed with Boston Carpal Tunnel Questionnaire, hand grip strength will be measured with dynamometer. Patient hand diagram will be marked according to patient's sensory symptoms. Median nerve cross-sectional area measurement at pisiform level with ultrasound, distal motor latency and sensory nerve conduction velocity with emg will be performed and recorded. Median nerve stiffness will be assessed with real-time elastography.

SUMMARY:
The aim of the study is to evaluate the prevalence of bifid median nerve in patients diagnosed with carpal tunnel syndrome (CTS) and whether it has a higher prevalence in CTS patients than in asymptomatic individuals, and to evaluate the characteristics of the bifid median nerve found and whether median nerve variations are predisposing factors in the development of CTS.

DETAILED DESCRIPTION:
Patients diagnosed with carpal tunnel syndrome electrophysiologically who applied to Etlik City Hospital physical therapy outpatient clinic will be included in the study.There are no sensitive groups.The research period was determined as 1 year.The sample size was done using G Power 3.1.9.4 statistical power analysis program for Windows.Based on the study conducted by Walker FO et al., the number of patients that would provide a significant difference (with a margin of error of 5% Type 1 and 20% Type 2, a study power of 80% and a confidence interval of 95%) was found to be 129 patients in total.Demographic and clinical characteristics of patients who meet the inclusion criteria and fill out the "Informed Consent Forum" will be recorded.General pain of the patients will be evaluated with the Visual Analogue Scale (Global Pain), symptom severity and functional status will be evaluated with the Boston Carpal Tunnel Questionnaire, and hand grip strength measurement will be evaluated with a dynamometer.The patient hand diagram will be marked according to the patient's sensory symptoms.Median nerve cross-sectional area will be measured at the pisiform level with ultrasound, and distal motor latency and sensory nerve conduction velocity will be measured with EMG and recorded.Median nerve stiffness will be evaluated by real-time elastography.

ELIGIBILITY:
Inclusion Criteria:

* Having typical Carpal Tunnel Sydnrome symptoms lasting longer than 3 months
* Carpal tunnel syndrome diagnosed with EMG
* Being a male/female >18 years of age

Exclusion Criteria:

* History of polyneuropathy, brachial plexopathy, thoracic outlet syndrome, or surgery in the wrist area
* Presence of inflammatory arthritis, hypothyroidism, pregnancy, rheumatological disorders, diabetes mellitus
* Presence of peripheral vascular disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 129 patients
Sampling Method: Non-Probability Sample
Enrollment: 129 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale(VAS) | This evaluation will be made and recorded at the beginning
  The VAS used for pain assessment consists of a line drawn in the form of a ruler,and numbers from 0 to 10(with 0 as ''no pain'' and 10 as ''unbearable pain'') were asked to score.

SECONDARY OUTCOMES:
Boston Carpal Tunnel Questionnaire | This evaluation will be made and recorded at the beginning.
  symptom severity and functional status scale
Dynamometer | This evaluation will be made and recorded at the beginning.
  Hand grip strength measurement test
Ultrasound | This evaluation will be made and recorded at the beginning.
  Median nerve cross-sectional area measurement at the pisiform level.
Real-time elastography. | This evaluation will be made and recorded at the beginning.
  Median nerve stiffness will be evaluated by real-time strain/sheer elastography.

CONTACTS AND LOCATIONS:
Overall Officials: Başak MANSIZ KAPLAN, assoc. prof., Study Chair — Ankara Etlik City Hospital; Ebru KARACA UMAY, prof. dr., Study Chair — Ankara Etlik City Hospital; Ajda BAL, prof. dr., Study Chair — Ankara Etlik City Hospital; Selin ÇELEBİER, assistant dr, Study Chair — Ankara Etlik Şehir Hastanesi
Locations (1):
- Etlik City Hospital, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bayrak IK, Bayrak AO, Kale M, Turker H, Diren B. Bifid median nerve in patients with carpal tunnel syndrome. J Ultrasound Med. 2008 Aug;27(8):1129-36. doi: 10.7863/jum.2008.27.8.1129. PMID 18645070
- [Background] Theofilopoulou S, Katouni K, Papadopoulos V, Pappas N, Antonopoulos I, Giavopoulos P, Chrysikos D, Filippou D. Variations of the Median Nerve and Carpal Tunnel Syndrome: a Systematic Review of the Literature. Maedica (Bucur). 2023 Dec;18(4):699-704. doi: 10.26574/maedica.2023.18.4.699. PMID 38348062
- [Background] Granata G, Caliandro P, Pazzaglia C, Minciotti I, Russo G, Martinoli C, Padua L. Prevalence of bifid median nerve at wrist assessed through ultrasound. Neurol Sci. 2011 Aug;32(4):615-8. doi: 10.1007/s10072-011-0582-8. Epub 2011 Apr 30. PMID 21533564